CLINICAL TRIAL: NCT05384587
Title: A Phase II Multicenter, Open-label, Single-arm Dose Escalation Study of Asciminib Monotherapy in 2nd and 1st Line Chronic Phase - Chronic Myelogenous Leukemia (ASC2ESCALATE)
Brief Title: Asciminib Monotherapy, With Dose Escalation, for 2nd and 1st Line Chronic Myelogenous Leukemia
Acronym: ASC2ESCALATE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABL001AUS08
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Chronic Myelogenous Leukemia - Chronic Phase
Keywords: CML; Chronic Phase; Asciminib; ASC2ESCALATE; T315I mutation; BCR-ABL; MMR; TKI; Tyrosine Kinase Inhibitor; molecular response; adult
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — asciminib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Asciminib (Experimental): 80 mg initial oral dose taken once a day with possible dose escalation
  Interventions: Drug: asciminib

INTERVENTIONS:
Drug: asciminib — Supplied in 40 mg and 100 mg tablets for oral use to be taken daily. Dose may be increased at 6 and 12 months based on molecular response with BCR-ABL1 Polymerase Chain Reaction testing.
  Other Names: ABL001

SUMMARY:
This will be a multicenter Phase II open-label study of asciminib in CML-CP patients who have been previously treated with one prior ATP- binding site TKI with discontinuation due to treatment failure, warning or intolerance. (2L patient cohort). In addition, newly diagnosed CML-CP patients who may have received up to 4 weeks of prior TKI are included in a separate 1L patient cohort.

DETAILED DESCRIPTION:
This trial consists of three periods: screening and baseline for up to 28 days, active treatment for up to 156 weeks and a safety follow up period for 30 days.

Ninety-two (92) 2L patients with CML-CP without T315I mutation who had 1 prior ATP-binding site TKI discontinued due to treatment failure, warning or intolerance will be considered for the current study. Patients will be tested at screening for the T315I mutation and excluded if the mutation is found.

To gain additional insights into the effect of asciminib in the 1L setting, an additional cohort of newly diagnosed CML-CP patients will be enrolled in the study. Based on the number of participating sites, it is approximated that between 60 and 90 patients could be enrolled. Enrollment of the 1L cohort will be stopped when a maximum of 90 patients have been enrolled or when approximately 60 patients have been enrolled and the 2L cohort is fully recruited, whichever comes first.

Informed consent will be obtained before any procedures are performed for the study including eligibility assessments.

All eligible patients will be initially treated with asciminib at 80 mg QD. At 6 months of study treatment, patients who have achieved BCR-ABL1IS ≤1% will continue on the same dose whereas those who have not will increase dose to 200mg QD.

At 12 months of study treatment, patients will be evaluated for the primary endpoint of the study (MMR at 12 month in 2L patient cohort) and will pursue one of the following:

* Continue on the current dose of asciminib if MMR is achieved
* Increase dose to 200 mg QD if on 80 mg QD dosing and MMR is not achieved
* Increase dose to 200 mg BID if on 200 mg QD dosing and MMR is not achieved
* Take the patient off the study and switch to Investigator's agent of choice if MMR is not achieved and it is in the interest of the patient based on investigator's clinical judgment of prospect treatment benefit.

ELIGIBILITY:
Key Inclusion Criteria:

Participants eligible for inclusion in this study must meet the following criteria: Criteria #1-5 are common to both patient cohorts (2L and 1L):

1. Signed informed consent must be obtained prior to participation in the study
2. CML-CP, no previous AP or BC
3. ≥ 18 years of age
4. ECOG performance status of 0, 1 or 2
5. Adequate end organ function within 14 days before the first dose of asciminib treatment.

   Patients with mild to moderate renal and hepatic impairment are eligible if:
   * Total bilirubin ≤ 3.0 x ULN without AST/ALT increase
   * Aspartate transaminase (AST) ≤ 5.0 x ULN
   * Alanine transaminase (ALT) ≤ 5.0 x ULN
   * Serum lipase ≤ 1.5 x ULN. For serum lipase > ULN and ≤ 1.5 x ULN, value should be considered not clinically significant and not associated with risk factors for acute pancreatitis
   * Alkaline phosphatase ≤ 2.5 x ULN
   * Creatinine clearance ≥ 30 mL/min as calculated using Cockcroft- Gault formula

   Criteria #6 and 7 are specific to the 2L patient cohort. These are meant to be either/or. It is not required to have both criteria satisfied.
6. Warning or failure (according to 2020 ELN Recommendations; Hochhaus et al) to 1L TKI therapy at the time of screening

   a. Warning is defined as: i. Six months after the initiation of treatment: BCR::ABL1IS >1-10% ii. Twelve months after the initiation of treatment: BCR::ABL1IS >0.1-1% b. Treatment failure/resistance to 1L TKI is defined as: i. BCR::ABL1IS >10% if 1L treatment duration between 6 and 12 months ii. BCR::ABL1IS >1% if 1L treatment longer than 12 months treatment iii. Beyond 12 months after initiation of treatment: loss of MMR
7. Treatment intolerance to 1L TKI,

   1. BCR::ABL1IS > 0.1% at screening
   2. Intolerance is defined as:

   i. Non-hematologic intolerance: Patients with grade 3 or 4 toxicity while on therapy, or with persistent grade 2 toxicity, unresponsive to optimal management, including dose adjustments (unless dose reduction is not considered in the best interest of the patient if response is already suboptimal) ii. Hematologic intolerance: Patients with grade 3 or 4 toxicity (absolute neutrophil count [ANC] or platelets) while on therapy that is recurrent after dose reduction to the lowest doses recommended by manufacturer

   Criteria #8 is specific to the 1L patient cohort
8. Patients with newly diagnosed CML-CP (treatment with a prior TKI (imatinib, or nilotinib, or dasatinib or bosutinib) for ≤ 4 weeks is allowed)

Key Exclusion Criteria:

1. Previous treatment

   1. With 2 or more ATP-binding site TKIs (for 2L patient cohort)
   2. More than 4 weeks with 1-ATP-binding site TKIs (for 1L patient cohort)
2. Previous treatment with asciminib
3. Known presence of the T315I mutation at any time prior to study entry
4. Known second chronic phase of CML after previous progression to AP/BC
5. Previous treatment with a hematopoietic stem-cell transplantation
6. Patient planning to undergo allogeneic hematopoietic stem cell transplantation
7. Cardiac or cardiac repolarization abnormality, including any of the following:

   * History within 6 months prior to starting study treatment of myocardial infarction (MI), angina pectoris, coronary artery bypass graft (CABG)
   * Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g., bifascicular block, Mobitz type II and third degree AV block)
   * QTcF at screening ≥450 msec (male patients), ≥450 msec (female patients)
   * Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:
   * Risk factors for Torsades de Pointes (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia
   * Concomitant medication(s) with a "Known risk of Torsades de Pointes" per www.crediblemeds.org that cannot be discontinued or replaced 7 days prior to starting study drug by safe alternative medication
   * Inability to determine the QTcF interval
8. History of acute pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis
9. Participation in a prior investigational study within 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever is longer
10. Treatment with medications that meet one of the following criteria is not allowed and should be switched to an alternative at least one week prior to the start of treatment with study treatment:

    * Strong inducers of CYP3A for patients on the dose of 80 mg QD and 200mg QD
    * Strong inducers and inhibitors of CYP3A for patients on the dose of 200 mg BID
11. Pregnant or nursing (lactating) women
12. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception. Highly effective contraception for women should be maintained throughout the study and for at least 7 days after the last dose.
13. Sexually active males unwilling to use a condom during intercourse while taking study treatment and for 7 days after stopping study (only for patients treated with asciminib).
14. Severe and/or uncontrolled concurrent medical disease that in the opinion of the Investigator could cause unacceptable safety risks or compromise compliance with the protocol (e.g. uncontrolled diabetes, active or uncontrolled infection; uncontrolled arterial or pulmonary hypertension, uncontrolled clinically significant hyperlipidemia).
15. History of other active malignancy within 3 years prior to study entry with the exception of previous or concomitant basal cell skin cancer and previous carcinoma in situ treated curatively.
16. Known hypersensitivity to the study treatment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2027-10-17 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who achieve Major Molecular Response (MMR) in the 2L setting | Baseline up to 12 months
  MMR is defined as BCR::ABL1IS ≤ 0.1%. A patient will be counted as having achieved MMR at 12 month if he/she meets the MMR criterion at 12 month.

SECONDARY OUTCOMES:
Percentage of participants achieving Molecular Response 4.5 (MR4.5) at 24 and 36 months | Baseline, 24 and 36 months
  Percentage of participants who achieve MR4.5 (defined as a ≥ 4.5 log reduction in BCR::ABL1 transcripts compared to the standardized baseline equivalent to ≤ 0.0032% BCR::ABL1/ABL % by international scale as measured by real time Polymerase Chain Reaction [PCR]) at the specified visits, i.e., if a patient achieves an MR4.5 but then loses it before or at the visit, he/she will be considered as non-responder for MR4.5 at that time point.
MMR Rate at visit (other than 12 month) | Baseline, 3, 6, 18, 24, 30 and 36 months
  Percentage of participants who achieve MMR (defined as BCR::ABL1IS ≤ 0.1%) at the specified visit, i.e., if a patient achieves an MMR earlier but then loses it at the visit, he/she will be considered as non-responder for MMR at the specified visit
MR2 Rate at visit | Baseline, 3, 6, 12, 18, 24, 30 and 36 months
  Percentage of participants who achieve MR2 (defined as a ≥ 2 log reduction in BCR::ABL1 transcripts) at the specified visit, i.e., if a patient achieves an MR2 earlier but then loses it at the visit, he/she will be considered as non-responder for MR2 at the specified visit
MR4 Rate at visit | Baseline, 3, 6, 12, 18, 24, 30 and 36 months
  Percentage of participants who achieve MR4 (defined as a ≥ 4 log reduction in BCR::ABL1 transcripts) at the specified visit, i.e if a patient achieves an MR4 earlier, but then loses it at the visit, he/she will be considered as non-responder for MR4 at the specified visit
MR4.5 Rate at visit | Baseline, 3, 6, 12, 18 and 30 months
  Percentage of participants who achieve MR4.5 (defined as a ≥ 4.5 log reduction in BCR::ABL1 transcripts) at the specified visit, i.e if a patient achieves an MR4.5 earlier, but then loses it at the visit, he/she will be considered as non-responder for MR4.5 at the specified visit
MMR Rate by visit | Baseline up to 3, 6, 12, 18, 24, 30 and 36 months
  Percentage of participants who achieve MMR at or before the specified visit, i.e., if a patient achieves an MMR but then loses it before or at the visit, he/she will still be considered as achieving MMR by that time point.
MR2 Rate by visit | Baseline up to 3, 6, 12, 18, 24, 30 and 36 months
  Percentage of participants who achieve MR2 (defined as a ≥ 2 log reduction in BCR::ABL1 transcripts) at or before the specified visit, i.e., if a patient achieves an MR2 but then loses it before or at the visit, he/she will still be considered as achieving MR2 by that time point.
MR4 Rate by visit | Baseline up to 3, 6, 12, 18, 24, 30 and 36 months
  Percentage of participants who achieve MR4 (defined as a ≥ 4 log reduction in BCR::ABL1 transcripts) at or before the specified visit, i.e., if a patient achieves an MR4 but then loses it before or at the visit, he/she will still be considered as achieving MR4 by that time point.
MR4.5 Rate by visit | Baseline up to 3, 6, 12, 18, 24, 30 and 36 months
  Percentage of participants who achieve MR4.5 (defined as a ≥ 4.5 log reduction in BCR::ABL1 transcripts) at or before the specified visit, i.e., if a patient achieves an MR4.5 but then loses it before or at the visit, he/she will still be considered as achieving MR4.5 by that time point.
Time to MMR | Baseline up to 36 months
  Time to MMR is defined and calculated as date of first documented MMR - start date of study treatment +1 day.
Duration of MMR | Baseline up to 36 months
  Duration of MMR is defined as the time from the date of first documented MMR to the earliest date of loss of MMR, progression to Accelerated Phase (AP) or Blast Crisis (BC), or CML-related death.
Time to Treatment Failure (TTF) | Baseline up to 36 months
  Time to treatment failure (TTF) is defined as the time from date of randomization to an event of treatment failure.
Progression Free Survival (PFS) | Baseline up to 36 months
  Time from the first dose of study treatment to the earliest occurrence of documented progression to Accelerated Phase (AP) or Blast Crisis (BC) or the date of death from any cause, before the end of the treatment phase.
Overall Survival (OS) | Baseline up to 36 months.
  Time from the first dose of study treatment to death due to any cause during the study.
Number of Adverse Events and Serious Adverse Events | Baseline up to 36 months
  Clinically significant findings for vitals, laboratory values and electrocardiogram (ECG) will be reported as adverse events and or serious adverse events as determined by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (80):
- United States (80):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Alaska Oncology and Hematology, Anchorage, Alaska
  - City of Hope Phoenix, Scottsdale, Arizona
  - USO Arizona Oncology, Tucson, Arizona
  - Onco Inst of Hope and Innovation, Cerritos, California
  - City of Hope National Medical, Duarte, California
  - UCSF Fresno Internal Medicine, Fresno, California
  - Virginia K Crosson Cancer Center, Fullerton, California
  - UCLA, Los Angeles, California
  - Alta Bates Summit Medical Center, Oakland, California
  - Lundquist Inst BioMed at Harbor, Torrance, California
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - The Stamford Hospital, Stamford, Connecticut
  - Florida Cancer Specialists, Fort Myers, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Florida Cancer Specialists-North, St. Petersburg, Florida
  - Florida Cancer Specialists East, Stuart, Florida
  - City Of Hope Atlanta, Atlanta, Georgia
  - Emory University School of Medicine Winship Cancer Institute, Atlanta, Georgia
  - Augusta University Georgia, Augusta, Georgia
  - Northwest Georgia Oncology Center, Marietta, Georgia
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Investigative Clinicl Rsrch of Indi, Indianapolis, Indiana
  - Holden Comp Can Cent Quad Cities U, Iowa City, Iowa
  - Wichita Community Clcl Onco Program, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Louisiana State University, Shreveport, Louisiana
  - Dana Farber Cancer Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Jackson Onc Associates, Jackson, Mississippi
  - University Missouri Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center, St Louis, Missouri
  - St Vincent Frontier Cancer Center, Billings, Montana
  - Nebraska Hematology Oncology P C, Lincoln, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Care Access Research Clifton, Clifton, New Jersey
  - Hackensack Meridian Health, Edison, New Jersey
  - Hackensack University Medical Ctr, Hackensack, New Jersey
  - Rutgers Cancer Institute of NJ, New Brunswick, New Jersey
  - UNM, Albuquerque, New Mexico
  - Clinical Research Alliance, Lake Success, New York
  - NYU Langone Long Island, Mineola, New York
  - Manhattan Hematol Oncol Associates, New York, New York
  - Mt Sinai Medical Center, New York, New York
  - New York Bld And Cancer Specialists, Port Jefferson, New York
  - SUNY Stony Brook Medical Oncology, Stony Brook, New York
  - SUNY Upstate Medical Center, Syracuse, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Novant Health Heart Vas Inst, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Uni Health Sci, Winston-Salem, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Hematology Oncology Care, Cincinnati, Ohio
  - James Cancer Hospital and Solove Research Institute Ohio State, Columbus, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Care Access Research, Easton, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Bon Secours Cancer Center, Greenville, South Carolina
  - Avera Cancer, Sioux Falls, South Dakota
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology P A, Austin, Texas
  - Texas Oncology, Dallas, Texas
  - Ctr For Cancer And Blood Disorders, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Univ of TX MD Anderson Cancer Cntr, Houston, Texas
  - Mays Cancer Center, San Antonio, Texas
  - Texas Oncology San Antonio, San Antonio, Texas
  - Texas Oncology Northeast Texas, Tyler, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Cancer Specialists, Gainesville, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VA Puget Sound Health Care System, Seattle, Washington
  - Fred Hutch Cancer Research, Seattle, Washington
  - Northwest Medical Specialties, Tacoma, Washington
  - Dean Health System, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Atallah EL, Mauro MJ, Sasaki K, Levy MY, Koller P, Yang D, Laine D, Sabo J, Gu E, Cortes JE. Dose-escalation of second-line and first-line asciminib in chronic myeloid leukemia in chronic phase: the ASC2ESCALATE Phase II trial. Future Oncol. 2024;20(38):3065-3075. doi: 10.1080/14796694.2024.2402680. Epub 2024 Oct 10. PMID 39387441